CLINICAL TRIAL: NCT03400774
Title: The Acute Effect of Moderate Intensity Stair-Climbing on Postprandial Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Jochen Kressler, Dr. Jochen Kressler, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2360098
Record Dates: First submitted 2017-12-14; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Postprandial Hyperglycemia
MeSH Terms: conditions — Hyperglycemia | interventions — Stair Climbing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Other): Oral glucose tolerance test with no stair-climbing
  Interventions: Other: Stair-climbing
- 1 minute (Experimental): Oral glucose tolerance test with 1 minute of stair-climbing
  Interventions: Other: Stair-climbing
- 3 minutes (Experimental): Oral glucose tolerance test with 3 minutes stair-climbing
  Interventions: Other: Stair-climbing
- 10 minutes (Active Comparator): Oral glucose tolerance test with 10 minutes stair-climbing
  Interventions: Other: Stair-climbing

INTERVENTIONS:
Other: Stair-climbing — Short bouts of moderate intensity stair-climbing

SUMMARY:
This study aims to investigate the effect of moderate intensity stair-climbing bouts of various durations on postprandial blood glucose. Participants will perform a standard oral glucose tolerance test (OGTT) using 75g of dextrose and with fingerstick blood glucose measurements at baseline and every 15 minutes after consuming the drink for one hour. On separate subsequent visits, participants will perform the same OGTT combined with three stair-climbing bouts lasting 1, 3, and 10 minutes starting 27, 25, and 18 minutes respectively after finishing the drink. Participants performed maximal aerobic capacity (VO2max) using a ramp treadmill test in order to assess the relative intensity of each stairclimbing trial.

ELIGIBILITY:
Inclusion Criteria:

* Defined as low risk per the American College of Sports Medicine (ACSM, Guidelines for Exercise Testing & Exercise Prescription, 20014 pg 30)
* Physical Activity Recall Questionnaire (PAR-Q) screening

Exclusion Criteria:

* Glucose intolerance
* Diabetes

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
Postprandial Blood Glucose | 1 hour
  Postprandial blood glucose after various durations of stair-climbing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bartholomae EM, Moore J, Ward K, Kressler J. Sex differences in postprandial glucose response to short bouts of exercise: A randomized controlled trial. J Sci Med Sport. 2019 Feb;22(2):181-185. doi: 10.1016/j.jsams.2018.07.009. Epub 2018 Jul 20. PMID 30077599

DOCUMENTS (3):
  • Informed Consent Form (2016-02-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT03400774/ICF_000.pdf
  • Statistical Analysis Plan (2016-02-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT03400774/SAP_001.pdf
  • Study Protocol (2016-02-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT03400774/Prot_002.pdf